CLINICAL TRIAL: NCT02782377
Title: Evaluation of the Rectal Reflex Using Anal Acoustic Reflectometry
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016GA002
Record Dates: First submitted 2016-03-21; First posted 2016-05-25 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Pelvic Floor Dysfunction
Keywords: Faecal Incontinence; Obstructive Defaecation; Rectal Prolapse
MeSH Terms: conditions — Encopresis; Rectal Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pelvic Floor Dysfunction: Observational study where patients with pelvic floor dysfunction undergo three AAR measurements. One at baseline, one with the catheter alongside and a third with the rectal balloon inflated. No intervention is performed
  Note, that initial inclusion of Squeeze parameters was detailed in error, these were not compared in this study and were compared in previous study

SUMMARY:
Anal Acoustic Reflectometry (AAR) is a reliable and reproducible technique that has been studied in our department over the last 6 years. Sound waves pass into a balloon placed in the anal canal and are used to measure the cross-sectional area. By gradually increasing and decreasing the pressure in the balloon the investigators can measure the pressure at which the cross-sectional area starts to increase and decrease, and the anal canal starts to open and close. This assessment mimics the natural opening and closing of the anal canal and the effect of squeezing the muscles.

The gold standard investigation of the anal sphincter muscles has been manometry which measures anal canal pressure at rest and during squeeze. However, it has limitations. In previous studies AAR has shown promise in the assessment of faecal incontinence and, that unlike manometry, it has been able to distinguish between different types of incontinence.

The Recto-anal Inhibitory Reflex (RAIR) is a normal response when the rectum fills with faeces, fluid or air, whereby there is a change in the pressures within the anal canal to determine the type of contents. This can be absent or altered in patients who have difficulty in opening their bowels. The RAIR is currently measured by anal manometry using a 4.9mm catheter, resulting in an anal canal which is already partially opened prior to the measurement, and potentially distorted.

AAR is considered a catheter free technique as the balloon has a cross-sectional area of only 0.4mm2 when collapsed. The investigators propose to measure the RAIR using a 1.7mm diameter catheter alongside the AAR balloon to determine the effect that its placement has on the recorded parameters of AAR. This aims to improve our understanding of the opening and closing of the anal canal in response to distension of the rectum.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 18 years old
2. Have capacity to consent to the study
3. Patients with pelvic floor dysfunction.

Exclusion Criteria:

1. Minors under the age of 18 years old
2. Patients who lack capacity to consent
3. Patients with known rectal tumours and proctitis
4. Asymptomatic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the pelvic floor clinic and neurogastroenterology with symptoms of pelvic floor dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Telford, MBChBMDFRCS, Study Chair — University Hospital of South Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klarskov N, Saaby ML, Lose G. A faster urethral pressure reflectometry technique for evaluating the squeezing function. Scand J Urol. 2013 Dec;47(6):529-33. doi: 10.3109/21681805.2013.776629. Epub 2013 Mar 19. PMID 23506115
- [Background] Hornung BR, Mitchell PJ, Carlson GL, Klarskov N, Lose G, Kiff ES. Comparative study of anal acoustic reflectometry and anal manometry in the assessment of faecal incontinence. Br J Surg. 2012 Dec;99(12):1718-24. doi: 10.1002/bjs.8943. PMID 23132420
- [Background] Saaby ML, Klarskov N, Lose G. Urethral pressure reflectometry before and after tension-free vaginal tape. Neurourol Urodyn. 2012 Nov;31(8):1231-5. doi: 10.1002/nau.22239. Epub 2012 Mar 27. PMID 22457059
- [Background] Klarskov N. Urethral pressure reflectometry. A method for simultaneous measurements of pressure and cross-sectional area in the female urethra. Dan Med J. 2012 Mar;59(3):B4412. PMID 22381095
- [Background] Mitchell PJ, Klarskov N, Telford KJ, Hosker GL, Lose G, Kiff ES. Viscoelastic assessment of anal canal function using acoustic reflectometry: a clinically useful technique. Dis Colon Rectum. 2012 Feb;55(2):211-7. doi: 10.1097/DCR.0b013e31823b2499. PMID 22228166
- [Background] Mitchell PJ, Klarskov N, Telford KJ, Hosker GL, Lose G, Kiff ES. Anal acoustic reflectometry: a new reproducible technique providing physiological assessment of anal sphincter function. Dis Colon Rectum. 2011 Sep;54(9):1122-8. doi: 10.1097/DCR.0b013e318223fbcb. PMID 21825892
- [Background] Cheeney G, Nguyen M, Valestin J, Rao SS. Topographic and manometric characterization of the recto-anal inhibitory reflex. Neurogastroenterol Motil. 2012 Mar;24(3):e147-54. doi: 10.1111/j.1365-2982.2011.01857.x. Epub 2012 Jan 11. PMID 22235880
- [Derived] Heywood NA, Sharma A, Kiff ES, Klarskov N, Telford KJ. Placement of a fine-bore rectal balloon catheter in the anal canal does not affect anal sphincter pressures: improving our understanding of physiological function with anal acoustic reflectometry. Colorectal Dis. 2020 Nov;22(11):1626-1631. doi: 10.1111/codi.15300. Epub 2020 Aug 30. PMID 32770704
- [Derived] Heywood NA, Sharma A, Kiff ES, Klarskov N, Telford KJ. A novel method for measurement of the recto-anal inhibitory reflex using anal acoustic reflectometry. Colorectal Dis. 2020 Nov;22(11):1632-1641. doi: 10.1111/codi.15110. Epub 2020 Sep 23. PMID 32367609

RESULTS

PARTICIPANT FLOW:
Groups:
- Pelvic Floor Dysfunction: Observational study where patients with pelvic floor dysfunction undergo three AAR measurements. One at baseline, one with the catheter alongside and a third with the rectal balloon inflated. No intervention is performed
Period: Overall Study
Arm/Group | Pelvic Floor Dysfunction
Started | 40
Completed | 35 (data from five of the patients were excluded due to interpretation difficulties)
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pelvic Floor Dysfunction
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 57.5 [34 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32

OUTCOME MEASURES:

1. Primary Outcome: Opening Pressure
Description: Measurements of differences in Opening pressure (Op - cm H2O) as measured by the AAR catheter.
  These measurements are taken at baseline with the rectal balloon collapsed (Pre-RAIR) and after inflation of 100mls air into rectal balloon (Post-RAIR).
Time Frame: during single study visit- measurement taken prior to balloon inflation and post balloon inflation
Measure: Median (Full Range); unit: cmH2O
Groups:
- Pre-Rair: AAR performed Prior to Rectal distension
- Post-RAIR: AAR performed after rectal distension
Arm/Group | Pre-Rair | Post-RAIR
Number analyzed (Participants) | 32 | 32
cmH2O | 34.44 [13.84 to 82.96] | 15.41 [0 to 50.53]

2. Primary Outcome: Opening Elastance
Description: Measurements of differences in Opening Elastance (Oe - cm H2O/mm2) as measured by the AAR catheter. These measurements are taken at baseline with the rectal balloon collapsed (Pre-RAIR) and after inflation of 100mls air into rectal balloon (Post-RAIR).
Time Frame: during single study visit- measurement taken prior to balloon inflation and post balloon inflation
Measure: Median (Full Range); unit: cmH2O/mm2
Arm/Group | Pre-Rair | Post-RAIR
Number analyzed (Participants) | 32 | 32
cmH2O/mm2 | 1.39 [0.74 to 2.18] | 1.1 [0 to 2.13]

3. Primary Outcome: Closing Pressure
Description: Measurements of differences in Closing Pressure (Cp - cm H2O) as measured by the AAR catheter. These measurements are taken at baseline with the rectal balloon collapsed (Pre-RAIR) and after inflation of 100mls air into rectal balloon (Post-RAIR).
Time Frame: during single study visit- measurement taken prior to balloon inflation and post balloon inflation
Measure: Median (Full Range); unit: cmH2O
Arm/Group | Pre-Rair | Post-RAIR
Number analyzed (Participants) | 32 | 32
cmH2O | 20.06 [6.01 to 55.92] | 8.00 [0 to 35.41]

4. Primary Outcome: Closing Elastance
Description: Measurements of differences in Closing Elastance (Ce - cm H2O/mm2) as measured by the AAR catheter. These measurements are taken at baseline with the rectal balloon collapsed (Pre-RAIR) and after inflation of 100mls air into rectal balloon (Post-RAIR).
Time Frame: during single study visit- measurement taken prior to balloon inflation and post balloon inflation
Measure: Median (Full Range); unit: cmH2O/mm2
Arm/Group | Pre-Rair | Post-RAIR
Number analyzed (Participants) | 32 | 32
cmH2O/mm2 | 1.31 [0.64 to 2.29] | 1.13 [0 to 1.73]

5. Primary Outcome: Hysteresis
Description: Measurements of differences in Hysteresis (%) as measured by the AAR catheter. These measurements are taken at baseline with the rectal balloon collapsed (Pre-RAIR) and after inflation of 100mls air into rectal balloon (Post-RAIR).
  Hysteresis is the extent of energy expenditure during opening and closing of the anal canal and represents the difference between opening and closing pressure and is expressed as a percentage
Time Frame: during single study visit- measurement taken prior to balloon inflation and post balloon inflation
Measure: Median (Full Range); unit: percent
Arm/Group | Pre-Rair | Post-RAIR
Number analyzed (Participants) | 32 | 32
percent | 39.71 [26.2 to 56.86] | 39.9 [0 to 82.28]

ADVERSE EVENTS:
Arm/Group | Pelvic Floor Dysfunction
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes